CLINICAL TRIAL: NCT06709885
Title: HDAC Inhibitor Combination with Immunochemotherapy in the Neoadjuvant Treatment of PMMR Locally Advanced Colon Cancer: a Multicenter, Double-arm, Phase II Randomized Controlled Study
Brief Title: HDAC Inhibitor Combination with Chemoimmunotherapy in the Neoadjuvant Treatment of PMMR Locally Advanced Colon Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Southwest Hospital, China (Other); Xinqiao Hospital of Chongqing (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Chongqing Medical University (Other); Chongqing University Cancer Hospital (Other); Chongqing General Hospital (Other); Chongqing Traditional Chinese Medicine Hospital (Other); Chongqing Shapingba District People's Hospital (Unknown); Chongqing Seventh People's Hospital (Unknown); Chongqing Renji Hospital, University of Chinese Academy of Sciences (Other Government); The 13th People's Hospital of Chongqing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIUNITE-02
Record Dates: First submitted 2024-10-13; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-09

CONDITIONS: Colon Adenocarcinoma
Keywords: HDAC inhibitors; pMMR/MSS; neoadjuvant immunochemotherapy; Oxaliplatin; Capecitabine
MeSH Terms: conditions — Colonic Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; tislelizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chidamide + Tislelizumab + chemotherapy (CapeOX ) (Experimental): 4 cycles of combination therapy (q3w; Day1 Oxaliplatin, 130mg/m2, iv.gtt; tislelizumab, 200mg/m2 iv.gtt; Day1,4,8,11Chidamide 20 mg BIW,PO; Day1-Day14, capecitabine 850-1000mg/m2, BID, PO)
  Interventions: Drug: Chidamide + Tislelizumab + chemotherapy (CapeOX )
- Neoadjuvant chemotherapy (CapeOX) (Active Comparator): 4 cycles Capeex (q3w; Day1 Oxaliplatin, 130mg/m2, iv.gtt; Day1-Day14, capecitabine, 850-1000mg/m2, BID, PO. ）
  Interventions: Drug: CapeOX

INTERVENTIONS:
Drug: Chidamide + Tislelizumab + chemotherapy (CapeOX ) — Chidamide + Tislelizumab + chemotherapy (CapeOX regimen): 4 cycles of combination therapy (q3w; Day1 Oxaliplatin, 130mg/m2, iv.gtt; tislelizumab, 200mg/m2 iv.gtt; Day1,4,8,11Chidamide 20 mg BIW,PO; Day1-Day14, capecitabine 850-1000mg/m2, BID, PO) ；After completing the surgery, Post-operation 4 cycles of Capeox
  Arms: Chidamide + Tislelizumab + chemotherapy (CapeOX )
Drug: CapeOX — 4 cycles (q3w; Day1 Oxaliplatin, 130mg/m2, iv.gtt; Day1-Day14, capecitabine, 850-1000mg/m2, BID, PO. ） Post-operation 4 cycles of Capeox
  Arms: Neoadjuvant chemotherapy (CapeOX)

SUMMARY:
The purpose of this clinical trial is to learn the safety and efficacy of HDAC inhibitors in combination with neoadjuvant immunochemotherapy compared to neoadjuvant therapy in the treatment of locally advanced colon cancer.

The main questions it aims to answer are:

Can HDAC inhibitors combined with neoadjuvant immunochemotherapy improve the rate of pCR and complete resection in patients? Are HDAC inhibitors combined with neoadjuvant immunochemotherapy safe and reliable? Does the combination of HDAC inhibitors and neoadjuvant immunochemotherapy achieve a better long-term prognosis than neoadjuvant therapy?

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to voluntarily join this study
2. Patients with colon cancer who are assessed by abdominal contrast-enhanced CT/abdominopelvic MRI as high-risk T3 (tumor destroys muscle wall and extends to pericolonic fat, protruding more than 5 mm into adjacent mesenteric fat) or T4 (tumor penetrates the visceral peritoneal surface or directly invades or adheres to adjacent organs or structures).
3. Adenocarcinoma of the colon confirmed by histopathological examination.
4. At least 18 years old, male or female.
5. Uncomplicated primary tumors (Perforation ； obstruction and bleeding that cannot be relieved by intervention)
6. The lower edge of the tumor is more than 12cm away from the anus.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Adequate bone marrow, liver, renal, and coagulation function as assessed by the laboratory as required by the protocol
9. Have not received any anti-tumor therapy for cancer in the past, including radiotherapy, chemotherapy, surgery, etc.;

Exclusion Criteria:

1. History of previous allergy to monoclonal antibodies, any component of HDACi, and capecitabine;
2. Has received or is receiving any of the following treatments in the past:

   1. Received any treatment against the mechanism of action of tumor immunity, such as immunization, HDACi, etc.
   2. Immunosuppressive drugs, or systemic hormonal drugs within 2 weeks prior to the first use of the study drug to achieve immunosuppressive purposes
   3. Receipt of a live attenuated vaccine within 4 weeks prior to the first use of study drug;
   4. Major surgery or severe trauma within 4 weeks prior to the first use of study drug;
   5. Receipt of systemic non-specific immunomodulatory therapy within 2 weeks prior to the first dose; Have received Chinese herbal medicines or proprietary Chinese medicines with anti-tumor indications within 2 weeks before the first dose.
3. Has any active autoimmune disease or history of autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism,
4. dMMR/MSI-H;
5. Presence of cardiac clinical symptoms or diseases that are not well controlled,
6. Severe infection (CTCAE > grade 2) within 4 weeks prior to the first use of study drug, with active tuberculosis infection found by medical history or CT examination,
7. Presence of active hepatitis B, hepatitis C 8.5 years of diagnosis of other malignant tumors, (adequately treated basal cell carcinoma of the skin or squamous cell skin cancer or carcinoma in situ of the cervix, etc., can be considered for enrollment);

9. Pregnant or lactating females; 10. As judged by the investigator, there are other factors that may lead to forced termination of the study, such as other serious diseases (including mental illnesses) requiring concomitant treatment, alcoholism, drug abuse, family or social factors, and factors that may affect the safety or compliance of the subject.

11. Have a history of immunodeficiency, including a positive HIV test, or have other acquired or congenital immunodeficiency disorders, or have a history of organ transplantation or allogeneic bone marrow transplantation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
pCR | The pCR rate will be evaluated after surgery, an average of 12 weeks
  pCR was defined as the absence, from surgical samples, of malignant cells in the primary site and regional lymph nodes

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  Defined as the time from randomization to relapse or death, whichever occurred first.
Overall survival (OS) | 3 years
  Defined as the time from randomization to date of death due to any cause according to RECIST version 1.1 recorded in the time period between randomization and disease progression or death to any cause
MPR | From enrollment to 12 Weeks of treatment end
  After neoadjuvant therapy, the percentage of residual viable tumor cells in the tumor bed ≤ 10%. Regardless of whether there are viable tumor cells left in the lymph nodes
Curative resection | From enrollment to 12 Weeks of treatment end
  Curative resection defined as complete tumor resection with all margins being negative.
ORR | From enrollment to 12 Weeks of treatment end
  Objective response is defined as a complete response (CR) or response (PR) according to RECIST v1.1
Down-staging of primary tumors | From enrollment to 12 Weeks of treatment end
  Down-staging of the resected tumour as measured by histopathological tumour diameter and stage according to the TNM staging system of AJCC (7th version).
Postoperative complications | 3 years
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.
Grade 3-4 adverse effects rate | From date of randomization until the date of death from any cause, assessed up to 3 years
  Rate of chemotherapy andHDACI and immunotherapy related severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: fan Li, PhD, Study Chair — Third Military Medical University
Locations (1):
- Daping Hospital， Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Argiles G, Tabernero J, Labianca R, Hochhauser D, Salazar R, Iveson T, Laurent-Puig P, Quirke P, Yoshino T, Taieb J, Martinelli E, Arnold D; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Localised colon cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Oct;31(10):1291-1305. doi: 10.1016/j.annonc.2020.06.022. Epub 2020 Jul 20. No abstract available. PMID 32702383
- [Background] Morton D, Seymour M, Magill L, Handley K, Glasbey J, Glimelius B, Palmer A, Seligmann J, Laurberg S, Murakami K, West N, Quirke P, Gray R; FOxTROT Collaborative Group. Preoperative Chemotherapy for Operable Colon Cancer: Mature Results of an International Randomized Controlled Trial. J Clin Oncol. 2023 Mar 10;41(8):1541-1552. doi: 10.1200/JCO.22.00046. Epub 2023 Jan 19. PMID 36657089
- [Background] Hu H, Zhang J, Li Y, Wang X, Wang Z, Wang H, Kang L, Liu P, Lan P, Wu X, Zhen Y, Pei H, Huang Z, Zhang H, Chen W, Zeng Y, Lai J, Wei H, Huang X, Chen J, Chen J, Tao K, Xu Q, Peng X, Liang J, Cai G, Ding K, Ding Z, Hu M, Zhang W, Tang B, Hong C, Cao J, Huang Z, Cao W, Li F, Wang X, Wang C, Huang Y, Zhao Y, Cai Y, Ling J, Xie X, Wu Z, Shi L, Ling L, Liu H, Wang J, Huang M, Deng Y; OPTICAL study group. Neoadjuvant Chemotherapy With Oxaliplatin and Fluoropyrimidine Versus Upfront Surgery for Locally Advanced Colon Cancer: The Randomized, Phase III OPTICAL Trial. J Clin Oncol. 2024 Sep 1;42(25):2978-2988. doi: 10.1200/JCO.23.01889. Epub 2024 Apr 2. PMID 38564700
- [Background] Michael-Robinson JM, Biemer-Huttmann A, Purdie DM, Walsh MD, Simms LA, Biden KG, Young JP, Leggett BA, Jass JR, Radford-Smith GL. Tumour infiltrating lymphocytes and apoptosis are independent features in colorectal cancer stratified according to microsatellite instability status. Gut. 2001 Mar;48(3):360-6. doi: 10.1136/gut.48.3.360. PMID 11171826
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Jordaan G, Liao W, Sharma S. E-cadherin gene re-expression in chronic lymphocytic leukemia cells by HDAC inhibitors. BMC Cancer. 2013 Feb 25;13:88. doi: 10.1186/1471-2407-13-88. PMID 23432814
- [Background] Shankar E, Pandey M, Verma S, Abbas A, Candamo M, Kanwal R, Shukla S, MacLennan GT, Gupta S. Role of class I histone deacetylases in the regulation of maspin expression in prostate cancer. Mol Carcinog. 2020 Aug;59(8):955-966. doi: 10.1002/mc.23214. Epub 2020 May 11. PMID 32391971
- [Background] Xie Y, Tang P, Xing X, Zhao Y, Cao S, Liu S, Lu X, Zhong L. In situ exploring Chidamide, a histone deacetylase inhibitor, induces molecular changes of leukemic T-lymphocyte apoptosis using Raman spectroscopy. Spectrochim Acta A Mol Biomol Spectrosc. 2020 Nov 5;241:118669. doi: 10.1016/j.saa.2020.118669. Epub 2020 Jul 2. PMID 32653824
- [Background] Liu L, Chen B, Qin S, Li S, He X, Qiu S, Zhao W, Zhao H. A novel histone deacetylase inhibitor Chidamide induces apoptosis of human colon cancer cells. Biochem Biophys Res Commun. 2010 Feb 5;392(2):190-5. doi: 10.1016/j.bbrc.2010.01.011. Epub 2010 Jan 7. PMID 20060381
- [Background] Wang H, Liu YC, Zhu CY, Yan F, Wang MZ, Chen XS, Wang XK, Pang BX, Li YH, Liu DH, Gao CJ, Liu SJ, Dou LP. Chidamide increases the sensitivity of refractory or relapsed acute myeloid leukemia cells to anthracyclines via regulation of the HDAC3 -AKT-P21-CDK2 signaling pathway. J Exp Clin Cancer Res. 2020 Dec 9;39(1):278. doi: 10.1186/s13046-020-01792-8. PMID 33298132
- [Background] Que Y, Zhang XL, Liu ZX, Zhao JJ, Pan QZ, Wen XZ, Xiao W, Xu BS, Hong DC, Guo TH, Shen LJ, Fan WJ, Chen HY, Weng DS, Xu HR, Zhou PH, Zhang YZ, Niu XH, Zhang X. Frequent amplification of HDAC genes and efficacy of HDAC inhibitor chidamide and PD-1 blockade combination in soft tissue sarcoma. J Immunother Cancer. 2021 Feb;9(2):e001696. doi: 10.1136/jitc-2020-001696. PMID 33637599
- [Background] Tu K, Yu Y, Wang Y, Yang T, Hu Q, Qin X, Tu J, Yang C, Kong L, Zhang Z. Combination of Chidamide-Mediated Epigenetic Modulation with Immunotherapy: Boosting Tumor Immunogenicity and Response to PD-1/PD-L1 Blockade. ACS Appl Mater Interfaces. 2021 Aug 25;13(33):39003-39017. doi: 10.1021/acsami.1c08290. Epub 2021 Aug 16. PMID 34433253
- [Background] He Y, Jiang D, Zhang K, Zhu Y, Zhang J, Wu X, Xia J, Zhu Y, Zou L, Hu J, Cui Y, Zhou W, Chen F. Chidamide, a subtype-selective histone deacetylase inhibitor, enhances Bortezomib effects in multiple myeloma therapy. J Cancer. 2021 Aug 27;12(20):6198-6208. doi: 10.7150/jca.61602. eCollection 2021. PMID 34539893
- [Background] Ding N, You A, Tian W, Gu L, Deng D. Chidamide increases the sensitivity of Non-small Cell Lung Cancer to Crizotinib by decreasing c-MET mRNA methylation. Int J Biol Sci. 2020 Jul 19;16(14):2595-2611. doi: 10.7150/ijbs.45886. eCollection 2020. PMID 32792859
- [Background] Liu L, Qiu S, Liu Y, Liu Z, Zheng Y, Su X, Chen B, Chen H. Chidamide and 5-flurouracil show a synergistic antitumor effect on human colon cancer xenografts in nude mice. Neoplasma. 2016;63(2):193-200. doi: 10.4149/203_150422N214. PMID 26774139